CLINICAL TRIAL: NCT01616641
Title: Orofacial Evaluation in Women With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, carmen paz santibanez hoyuela, orofacial evaluation in women with rheumatoid arthritis, Federal University of São Paulo
Other Study IDs: Orofacial
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; bite force; grip strenght; oral health; quality of life
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- rheumatoid arthritis group: 75 patients with rheumatoid arthritis
- control group: 75 healthy women

SUMMARY:
Rheumatoid arthritis (RA) can affect any synovial joint. Unlike the hand, ever so valued in the physical examination of patients with RA, the joints in the area of the jaw and neck may also be affected in this disease and have their involvement usually underdiagnosed. There are few studies evaluating the incidence of orofacial alteration in the examination as well as the correlation between bite force (BF) and clinical and functional parameters in these patients. The aim of our study was to chacacterize the orofacial alterations in RA patients, correlate the results of the orofacial evaluation with clinical and disease activity parameters, and correlate the bite force with the hand strenght.

ELIGIBILITY:
Inclusion Criteria:

RA group:

* rheumatoid arthritis (American College of Rheumatology)

Control group:

* healthy

Exclusion Criteria:

* edentate be total, have been subjected to surgical procedure in the last six months in the region of the hands or oral maxillo facial

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 150 individuals, half of them, 75 were rheumatoid arthritis and the others 75 consisted the group control
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-06; Study Completion 2012-06 (Actual)